CLINICAL TRIAL: NCT00819897
Title: Longitudinal Study in Clinical Isolated Syndrome Patients Treated With Interferon Beta. Correlation With Cognitive Disorders and Quality of Life.
Brief Title: Longitudinal Study in Clinically Isolated Syndrome (CIS) Patients Treated With Interferon Beta
Acronym: QUALICIS
Status: Terminated | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 08-PP-05
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Clinically Isolated Syndrome
Keywords: MS; CIS; IFN; MRI; OCT; QOL

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the role of cognitive disorders and quality of life in patients with CIS, considered as high risk to develop an MS, treated with interferon Beta. This prospective observational study will include 120 patients, all treated and evaluated annually with neurological extensive examination, ophthalmologic screening (OCT, OF, VEP, VF), auto questionnaire about fatigue (musicol, ELIF), quality of life (SEP-59), and conventional MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years,
* Patients with CIS and temporo spatial dissemination for less than one year
* Patient without prior immunomodulatory treatment
* Patient informed of CIS diagnosis and MS according to McDonald criteria,
* Patients with EDSS inferior or egal to 5,5
* Patients usually french-reader and with MMS >24
* Patients informed of study protocol
* Patients agree to sign informed consent
* Patients with affiliation number from social French département.

Exclusion Criteria:

* Secondary progressive MS
* Patient with acute relapse
* Patient already treated with IFN
* corticosteroids less than 15 days
* Patient with severe dépressive disorders
* Patient already included in clinical study
* Patient < 18 years
* Patient with known contra indications for beta interféron
* Every reason with can provoke an interruption of the study, regarding a patient empechment
* Contre indications for MRI or other tests required in the study
* pregnancy or lactation
* patient Under juridic protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with CIS and temporo spatial dissemination for less than one year without prior immunomodulatory treatment
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Clinical exams performed at Baseline and every year during 3 years Neurological examination: relapses recording and EDSS. Quality of life: SEP-59, MusiQOL. Neuropsychological screening | 3 years

SECONDARY OUTCOMES:
Fatigue test: MS Fatigue, MRI (T1 gadolinium, T2, sagittale T1, acquisition volumique 3D T1), Optical coherence tomography (OCT) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine LEBRUN-FRENAY, MDPH, Principal Investigator — University hospital of Nice
Locations (17):
- France (17):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - University hospital of Côte de Nacre, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Général de DIJON, Dijon
  - Hôpital Roger Salengro, Lille
  - Hôpital de Saint Philibert, Lomme
  - Centre Hospitalier de la Timone, Marseille
  - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU Nice, Nice
  - CHU de Montpellier-Nîmes - Hôpital Caremeau, Nîmes
  - Hôpital de Poissy, Poissy
  - CHU de Reims, Reims
  - Hôpital Pontchaillon, Rennes
  - CHRU de Strasbourg, Strasbourg
  - Hôpital Purpan, Toulouse